CLINICAL TRIAL: NCT04278625
Title: Pharmacokinetics of Acetaminophen in Pediatric Patients With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Peter Winch (Other)
Responsible Party: Sponsor-Investigator, Peter Winch, Associate Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00000766
Record Dates: First submitted 2020-02-10; First posted 2020-02-20 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-11

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cyanotic CHD: Cyanotic congenital heart disease (CHD) patients presenting for Fontan palliation.
  Interventions: Drug: Acetaminophen
- Acyanotic CHD: Acyanotic congenital heart disease (CHD) patients presenting for repair via median sternotomy.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — IV acetaminophen given as part of standard of care.

SUMMARY:
This is a prospective study of pediatric patients with congenital heart disease, in which acetaminophen serum concentrations will be measured following a single intraoperative intravenous dose of acetaminophen. These levels will be used to develop a pharmacokinetic model. Serum concentrations will be compared between two groups of patients: (1) cyanotic patients presenting for the Fontan completion operation and (2) patients with acyanotic congenital heart disease presenting for repair via median sternotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for Fontan palliation or for surgical repair requiring median sternotomy, will be included in the study.
* Only patients who receive intravenous acetaminophen in the operating room will have serum levels drawn.

Exclusion Criteria:

* Documentation of an allergy to acetaminophen
* Severe hepatic disease or other contraindications to acetaminophen use
* Patient has received acetaminophen within 24 hours of their procedure

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric congenital heard disease patients undergoing cardiac surgery and receiving IV acetaminophen during their surgical procedure as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyanotic CHD | Acyanotic CHD
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyanotic CHD | Acyanotic CHD | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.6 [3.12 to 4.1] | 3.58 [2.53 to 4.9] | 3.59 [2.06 to 6.31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 10 | 12 | 22
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Cardiopulmonary bypass time [Median (Inter-Quartile Range); unit: minutes] — The length of time the subjects were on cardiopulmonary bypass during the surgery.
  minutes | 78 [57.5 to 92] | 73 [44 to 84] | 73.5 [45.2 to 88]

OUTCOME MEASURES:

1. Primary Outcome: Acetaminophen Serum Concentrations
Description: The amount of acetaminophen in the blood stream at each time point after receiving a standard dose.
Time Frame: 15-20 minutes; 30-40 minutes; 50-70 minutes; 80-100 minutes; 2 Hours, 4 Hours; and 6-Hours Post-IV acetaminophen administration
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | Cyanotic CHD | Acyanotic CHD
Number analyzed (Participants) | 15 | 15
mcg/mL
  15-20 minutes | 19 [16 to 24] | 17 [15 to 19]
  30-40 minutes | 13 [12 to 15] | 13 [12 to 14]
  50-70 minutes | 11 [9.6 to 11] | 10 [9.2 to 11]
  80-100 minutes | 8.7 [8.3 to 9.5] | 8 [6.9 to 9.1]
  2 Hours | 6.9 [6.3 to 7.4] | 6.6 [5.3 to 8.4]
  4 Hours | 4.1 [3.3 to 4.7] | 2.9 [2.7 to 4.4]
  6 Hours | 2.5 [1.8 to 3.3] | 1.7 [1.4 to 2.9]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Cyanotic CHD | Acyanotic CHD
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT04278625/Prot_SAP_000.pdf